CLINICAL TRIAL: NCT06760338
Title: Factors Associated With Quality of Life in Patients With Knee Osteoarthritis
Brief Title: Factors Associated With Quality of Life in Knee Osteoarthritis
Status: Completed | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Emrah Afsar, Phd, Kutahya Health Sciences University
Other Study IDs: 2024-e
Record Dates: First submitted 2024-12-30; First posted 2025-01-06 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study was to investigate the relationship between quality of life and factors that may affect quality of life (pain, stiffness, functional status and depression) in knee osteoarthritis.

DETAILED DESCRIPTION:
Participants aged between 40-65 years, willing to participate in the study and diagnosed with knee osteoarthritis will be included in the study. Necessary demographic information will be obtained with the prepared data form. Numerical Rating Scale (NRS), Western Ontario and Mcmaster Universities Osteoarthritis Index (WOMAC Osteoarthritis Index), Knee Injury and Osteoarthritis Outcome Score (KOOS), Lower Extremity Functional Scale (LEFS), Beck Depression Scale, Short Form - 36 (Quality of Life Questionnaire) will be used for evaluation. The data obtained in the study will be entered into SPSS 17 package programme (Greasley, 2007). Minimum-maximum values, arithmetic mean and standard deviation will be used to evaluate numerical data, and frequency distributions and percentages will be used to summarise categorical data. The data of the study will be analysed using Analysis of Moment Structures (AMOS) statistical package programmes. In all analyses, p<0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Being diagnosed with knee osteoarthritis
* In studies between the ages of 40 and 65

Exclusion Criteria:

* Other orthopaedic surgery in the lower extremity
* Cognitive impairment at a level that prevents understanding and answering the questionnaire
* Presence of neurological disease

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include people aged between 40-65 years, who volunteered to participate in the study and diagnosed with knee osteoarthritis.
Sampling Method: Probability Sample
Enrollment: 174 (Actual)
Dates: Start 2025-01-06 (Actual); Primary Completion 2025-07-25 (Actual); Study Completion 2025-07-25 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale - NRS | 1 minute
  It is an 11-point scale with numbers from 0 to 10, with 0 indicating 'no pain' and 10 indicating 'the worst pain imaginable'. Patients are asked to choose a single number from the scale that best represents their level of pain.
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 3 minute
  WOMAC is a valid and reliable questionnaire that is frequently used in clinics and research in patients with knee OA. WOMAC is a self-administered assessment tool. It consists of 24 questions and three subcategories (pain, stiffness and physical function). Pain is assessed with 5 questions, stiffness with 2 questions and physical function with 17 questions. Each question is scored between 0-4 (0 = none, 1 = mild, 2 = moderate, 3 = severe, 4 = extreme). Subcategories are evaluated within themselves. The maximum score is: 20 points for pain, 8 points for stiffness and 68 points for physical function. High WOMAC scores indicate an increase in pain and stiffness and deterioration in physical function.
Knee Injury and Osteoarthritis Outcome Score (KOOS) | 5 minute
  It is a scale used to evaluate symptoms and functional status related to knee osteoarthritis. It consists of a total of 42 items and 5 subscales including pain, patient's views on other symptoms, activities of daily living, sports and recreational activities and knee-related quality of life. Each question is scored between 0 and 4 points. Each subscale is scored between 0-100 (0 indicates a serious problem and 100 indicates no problem).
Lower Extremity Functional Scale (LEFS) | 2 minute
  It is used to classify the functional status of individuals. LEFS is a 5-point Likert scale consisting of 20 questions with options (graded between 0 and 4 points). The total score ranges from 0-80. Higher scores represent a better functional status.
Beck Depression Scale | 5 minute
  The Beck Depression Scale is a self-report questionnaire that assesses the presence and severity of depressive symptoms. It consists of 21 items. Each item is scored on a four-point scale ranging from 0 (none) to 3 (severe). Total scores can vary between 0 and 63. The reliability and validity findings of the questionnaire adapted to Turkish have been obtained.
Short Form - 36 Quality of Life Questionnaire (SF-36) | 7 minute
  The Short Form - 36 Quality of Life Questionnaire (SF-36) is a general measure of health status, rather than measuring the outcomes of specific conditions. There is evidence that the SF-36 can be used to monitor musculoskeletal conditions. The SF-36 is a health-related quality of life questionnaire consisting of 8 scales (physical functioning, role limitations due to physical health problems, pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, mental health). Responses to items are converted into scale scores from 0 (worst health) to 100 (best health). One physical and one mental summary health measure are derived from the 8 scales.

CONTACTS AND LOCATIONS:
Overall Officials: Emrah Afsar, Phd, Principal Investigator — Kutahya Health Science University
Locations (1):
- Kutahya Health Science University, Kütahya, Turkey (Türkiye)